CLINICAL TRIAL: NCT04086095
Title: Feasibility Study - Neofact Feasibility Study of the Application Aid Neofact (Formerly: QuickSF) in the Less Invasive Surfactant Administration (LISA) in Premature Infants With Respiratory Distress Syndrome.
Brief Title: Feasibility Study - Neofact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Klinikum Stuttgart (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: feasibility study - Neofact
Record Dates: First submitted 2019-09-03; First posted 2019-09-11 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-08

CONDITIONS: Respiratory Distress Syndrome in Premature Infant; Surfactant Deficiency Syndrome Neonatal
Keywords: Respiratory Distress Syndrome; Less Invasive Surfactant Administration; Neofact; Preterm babies
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Premature babies with Respiratory Distress Syndrome and the medical need for surfactant administration (defined as FiO2 ≥ 0.3 or mod. Silverman Andersen Respiratory Severity Score ≥ 5) while treated with CPAP-support and in a gestational age >26+0 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Surfactant administration will be done via videolaryngoscopy and the application aid Neofact in neonates with respiratory distress syndrome and airway support with CPAP. Alveofact is used as Surfactant in its standard dosage of 100 mg / kg
  Interventions: Device: Neofact application aid

INTERVENTIONS:
Device: Neofact application aid — The Neofact application aid is a specifically for the LISA procedure designed guide of a soft catheter and replaces the Magill forceps. Catheter (3.5 Fr.) and guide are already combined and packed together sterile. The catheter tip is marked in black (1cm).

SUMMARY:
For therapy of respiratory distress syndrome (RDS) in premature babies, there are several established options. An important therapeutic aspect is the tracheal administration of exogenous surfactant into the child's lung.

In the recent years, several methods have been developed. The methods differ in the selected ventilation mode (intubation with mechanical ventilation vs. Continous Positive Airway Pressure (CPAP)-supported spontaneous breathing) and in the way in which the application of surfactant is technically conducted (via endotracheal tube, endotracheal catheter or nebulization).

In selection of ventilation technique, there is an upcoming trend towards less invasive respiratory support via CPAP. While this may increase the rate of complications on the one side (i.e. pneumothorax), it shows much lower oxygen demand and a shorter need for mechanical ventilation on the other side.

In the selection of the administration technique, different methods were repeatedly developed to adapt the surfactant administration to the CPAP therapy. In this study, a newly developed and in the European Community now certified (CE-Mark) application aid (Neofact) will be tested for the first time on preterm infants, to verify the feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with respiratory distress syndrome and the need for Surfactant administration (oxygen requirement with FiO2 ≥ 30% and/or mod. Silverman Andersen Respiratory Severity Score (RSS) ≥ 5)
* Respiratory support with non-invasive CPAP at the time of Surfactant administration

Exclusion Criteria:

* Preterms with an gestational age < 26+0 weeks
* Preterms with malformations of the respiratory tract
* Clinical decision on intubation / surfactant application via endotracheal tube e.g. because of respiratory drive disorder
* (Missing parental consent)
* (Attending physician is not delegated by the principal investigator)

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
feasibility of the application aid Neofact | Administration of surfactant + 30 minutes
  Feasibility will be defined as a correct intratracheal position of the catheter (visually controlled via videolaryngoscope) OR responsiveness of the child to the surfactant administration (defined as decrease of the fraction of inspired oxygen (FiO2) of at least 0.05 within 30 minutes after the application OR FiO2 decrease to 0.21 with simultaneous improvement of the modified Silverman Andersen Respiratory Severity Score (RSS) ≥ 2 within 30 minutes after the application) without switching to a conventional LISA method
  RSS in the modified version of McAdams RM et al. The RSS consists of 5 categories that assess the respiratory work of the child in a range from 0 to 2 in each category. This results in a summarized score of 0 to 10, in which 0 defines a healthy neonate without increased work of breathing and 10 a neonate with maximum respiratory distress.

SECONDARY OUTCOMES:
Duration of the surfactant administration procedure | up to 20 minutes
  Measured time from the beginning of the initial insertion of the laryngoscope (plate tip passes the lips) to the removal of the application aid Neofact (Neofact tip passes the lips).
Duration of the laryngoscopy | up to 15 minutes
  Measured time from the beginning of the initial insertion of the laryngoscope (plate tip passes the lips) to the removal of the laryngoscope (plate tip passes the lips).
Need for intubation and mechanical ventilation | 48 hours after administration
  Number of neonates that need intubation and mechanical ventilation in the observational period of 48 hours after surfactant administration
Number of attempts needed for the correct application | during application procedure
  to evaluate how good the handling of the application aid will be
Occurrence of complications | during application procedure
  Number of decreases of oxygen saturation (< 80% SpO2), bradycardia (< 80 / min), tachycardia (> 200 / min), arterial hypo- (middle arterial blood pressure < Gestational Age (GA)) or hypertension (middle arterial blood pressure > GA + 20), onset and / or severity of coughing, choking, apnea & laryngospasm during the procedure
Colonization of the catheter tip | up to 20 minutes
  Name of germs and their number of colony forming units (CFU) placed on the catheter tip. To evaluate if there is a risk of contamination

CONTACTS AND LOCATIONS:
Overall Officials: Christian A. Maiwald, Dr., Study Chair — Department of Neonatology
Locations (2):
- Germany (2):
  - Klinikum Stuttgart - Olgahospital, Stuttgart, Baden-Wurttemberg
  - University Hospital, Tübingen, Baden-Wurttemberg

REFERENCES:
- [Background] Lindner W, Vossbeck S, Hummler H, Pohlandt F. Delivery room management of extremely low birth weight infants: spontaneous breathing or intubation? Pediatrics. 1999 May;103(5 Pt 1):961-7. doi: 10.1542/peds.103.5.961. PMID 10224173
- [Background] Dani C, Bertini G, Pezzati M, Cecchi A, Caviglioli C, Rubaltelli FF. Early extubation and nasal continuous positive airway pressure after surfactant treatment for respiratory distress syndrome among preterm infants <30 weeks' gestation. Pediatrics. 2004 Jun;113(6):e560-3. doi: 10.1542/peds.113.6.e560. PMID 15173537
- [Background] Morley CJ, Davis PG, Doyle LW, Brion LP, Hascoet JM, Carlin JB; COIN Trial Investigators. Nasal CPAP or intubation at birth for very preterm infants. N Engl J Med. 2008 Feb 14;358(7):700-8. doi: 10.1056/NEJMoa072788. PMID 18272893
- [Background] Maiwald CA, Neuberger P, Vochem M, Poets C. QuickSF: A New Technique in Surfactant Administration. Neonatology. 2017;111(3):211-213. doi: 10.1159/000450823. Epub 2016 Nov 15. PMID 27842300
- [Background] McAdams RM, Hedstrom AB, DiBlasi RM, Mant JE, Nyonyintono J, Otai CD, Lester DA, Batra M. Implementation of Bubble CPAP in a Rural Ugandan Neonatal ICU. Respir Care. 2015 Mar;60(3):437-45. doi: 10.4187/respcare.03438. Epub 2014 Nov 11. PMID 25389349
- [Derived] Maiwald CA, Dick J, Marschal M, Gille C, Franz AR, Poets CF. Microbiological analyses of nasally guided catheters after less invasive surfactant administration - a pilot study. BMC Pediatr. 2020 May 19;20(1):234. doi: 10.1186/s12887-020-02147-0. PMID 32429874